CLINICAL TRIAL: NCT04061603
Title: iCLAS™ for Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-200
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Symptomatic persistent atrial fibrillation that failed at least one class I or Class III AAD with no prior history of ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- iCLAS Ablation (Experimental): Ablation of the left and right atrium with the Adagio Medical iCLAS System
  Interventions: Device: Adagio AF Cryoablation System (iCLAS™)

INTERVENTIONS:
Device: Adagio AF Cryoablation System (iCLAS™) — Endovascular ablation of the left and right atrium

SUMMARY:
Clinical study to evaluate the safety and efficacy of the Adagio AF Cryoablation System (iCLAS™) in the ablation treatment of symptomatic, persistent atrial fibrillation (PsAF). Data will be used to support a pre-market application (PMA)

DETAILED DESCRIPTION:
A staged pre-market, single-arm, clinical study designed to collect acute and long-term safety and efficacy data for the Adagio AF Cryoablation System (iCLAS™). Patient population will consist of symptomatic, persistent AF subjects completing a de novo ablation procedure. Enrollment will be 200 subjects at up to 20 global investigational sites. Subjects will receive an ablation with the ultra-low cryoablation device. Follow-up will include assessment at one, three, six, and twelve months.

ELIGIBILITY:
INCLUSION CRITERIA

IC1 Male or female between the ages of 18 and 80 years

IC2 Currently scheduled for an ablation of symptomatic, PsAF defined as continuous AF that is sustained > 7-days and ≤ 12 months and documented by the following: a. Physician's note indicating continuous AF > 7 days and ≤ 12 months, AND b. One of the following: i. 24-hour Holter within 180 days of enrollment showing continuous AF, OR ii. Two electrocardiograms from any forms of rhythm monitoring (e.g., 12-lead ECGs or single lead ECGs) completed ≥ 7 days apart within 180 days of enrollment.

IC3 Refractory to at least one class I or III AAD. (Refractory defined as not effective, not tolerated or not desired)

IC4 Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study

IC5 Willingness and ability to give an informed consent

EXCLUSION CRITERIA

EC 1 In the opinion of the Investigator, any known contraindication to an atrial ablation, TEE, or anticoagulation. Including, but not limited to, the identification of any atrial thrombus or evidence of sepsis

EC 2 Any duration of continuous AF lasting longer than 12-months

EC 3 History of previous left atrial ablation or surgical treatment for AF/AFL/AT

EC 4 Atrial fibrillation secondary to electrolyte imbalance, active thyroid disease, or any other reversible or non-cardiac cause

EC 5 Structural heart disease as described below:

1. Left ventricular ejection fraction (LVEF) < 40% based on most recent TTE
2. Left atrial size > 55 mm (parasternal long axis view) documented within 6-months of screening
3. NYHA Class III or IV heart failure documented within the previous 12-months
4. An implanted pacemaker or ICD
5. Previous cardiac surgery, ventriculotomy, or atriotomy (excluding atriotomy for CABG),
6. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve
7. Interatrial baffle, closure device, patch, or PFO occluder
8. Presence of a left atrial appendage occlusion device
9. Presence of any pulmonary vein stenting devices
10. Coronary artery bypass graft (CABG) or PTCA procedure within 6 months prior to procedure
11. Unstable angina or ongoing myocardial ischemia
12. Myocardial infarction within the previous six (6) months prior to procedure
13. Moderate or severe mitral insufficiency or stenosis based on most recent TTE
14. Atrial myxoma
15. Significant congential anomaly

EC 6 BMI > 40

* BMI >35 and no prior sponsor approval into the study

EC 7 Any previous history of cryoglobulinemia

EC 8 History of blood clotting or bleeding disease

EC 9 History of severe COPD requiring steroid use in the previous 12-months

EC 10 History of severe sleep apnea (AHI > 30) not currently treated with a CPAP machine or other mechanical device

EC 11 Any prior history of documented cerebral infarct including recent TIA (within one year) or systemic embolism (excluding a post-operative DVT)

EC 12 Any prior history or current evidence of hemidiaphragmatic paralysis

EC 13 Pregnant or lactating (current or anticipated during study follow-up)

EC 14 Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study

EC 15 Any other condition that, in the judgment of the investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center, COVID-19 related concerns)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of the proportion of subjects who are free from device/procedure related Major Adverse Events (MAEs) that occur following the cryoablation procedure. | 12-months
  MAEs include any of the following:
  * Death
  * Myocardial infarction
  * Cardiac perforation/pericardial tamponade
  * Cerebral infarct or systemic embolism
  * Major bleeding requiring transfusion of blood products
  * Mitral or tricuspid valve damage
  * Symptomatic pulmonary vein stenosis
  * Severe (≥ 70%) pulmonary vein stenosis
  * Permanent phrenic nerve injury
  * Access site complications requiring pharmacological or surgical intervention
  * Atrio-esophageal fistula
  * Pericarditis
  * Heart block requiring a permanent pacemaker
  * Vagal nerve injury with GI dysmotility
  * Other serious adverse device effects (SADEs), including TIAs, adjudicated by an independent Clinical Events Committee (CEC) as "probably or definitely related" to the Adagio System
Analysis of the proportion of subjects receiving a single cryoablation who are free from any documented left atrial arrhythmia (AF/AFL/AT). | 12-months
  The primary effectiveness endpoint will be based on a centralized core lab interpretation of the recordings used in the endpoint analysis.

SECONDARY OUTCOMES:
Recording and analysis of all identified SAEs and SADEs through 12-months post-procedure. | 12-months
  Events will be sub-stratified based on time to event as follows:
  * Early onset (procedure through 7-days post-ablation)
  * Peri-procedure (> 7-days through 30-days post-ablation)
  * Late onset (>30-days post ablation)
Analysis of the proportion of subjects with acute procedural (ablation) success | 20-minutes following last ablation
  Documentation of pulmonary vein isolation and posterior wall isolation

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — Valley Hospital
Locations (21):
- United States (16):
  - Grandview Medical Center, Birmingham, Alabama
  - Banner Health, Phoenix, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - University of California San Diego, San Diego, California
  - South Denver Cardiology Associates, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Prairie Heart Research Institute, Springfield, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Valley Hospital, Ridgewood, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Staten Island University Hospital - Northwell Health, Staten Island, New York
  - Ohio Health Research Institute, Columbus, Ohio
  - Baylor St. Luke's Medical Center, Houston, Texas
- Belgium (2):
  - Onze Lieve Vrouwziekenhuis, Aalst
  - ZNA Middelheim, Antwerp
- Southlake Regional Medical Centre, Newmarket, Ontario, Canada
- Netherlands (2):
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No